CLINICAL TRIAL: NCT07336628
Title: Propofol Versus Remifentanil for BIS-Guided Sedation in Gastroscopy: A Randomized Controlled Trial
Brief Title: BIS-Guided Propofol vs Remifentanil for Gastroscopy: Effects on Procedure Start Time and Recovery
Acronym: ROPOGAST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Cansu Ofluoğlu, Specialist in Anesthesiology and Reanimation, Fatih Sultan Mehmet Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: FSMTRHSEDO
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Conscious Sedation
Keywords: Procedural Sedation; Ramsay Sedation Scale; Awakening Time; Conscious Sedation; BIS Monitoring; Bispectral Index; Gastroscopy; Remifentanil; Propofol
MeSH Terms: interventions — Propofol; Remifentanil

STUDY DESIGN:
Intervention Model Description: Two-arm parallel design with 1:1 randomization. No crossover.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are sedated during the procedure and unaware of group assignment. Outcomes assessors (recovery room nurses, independent observers assessing Ramsay scores) are blinded to group allocation. The anesthesiologist administering sedation is necessarily unblinded to allow appropriate drug titration but does not participate in outcome assessment. Endoscopists are blinded to group allocation and BIS values.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol Group (Active Comparator): Patients receive midazolam 2 mg IV premedication followed by continuous propofol infusion (100-150 µg/kg/min) titrated to maintain BIS 60-80.
  Interventions: Drug: Propofol (Astra-Zeneca)
- Remifentanil Group (Active Comparator): Patients receive midazolam 2 mg IV premedication followed by remifentanil loading dose (1 µg/kg) and continuous infusion (0.025-0.1 µg/kg/min) titrated to maintain BIS 60-80.
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Propofol (Astra-Zeneca) — Continuous intravenous infusion of propofol at 100-150 µg/kg/min, titrated to maintain bispectral index (BIS) values between 60 and 80 and Ramsay Sedation Scale scores of 2-3. Infusion is initiated after endoscopy team confirms readiness and continued until procedure completion. Administered only to participants in the Propofol Group.
  Other Names: Propofol Injectable Emulsion
  Arms: Propofol Group
Drug: Remifentanil — Intravenous loading dose of remifentanil 1 µg/kg administered over 60 seconds, followed by continuous infusion at 0.025-0.1 µg/kg/min. Infusion rate is titrated to maintain bispectral index (BIS) values between 60 and 80 and Ramsay Sedation Scale scores of 2-3. Infusion is initiated after endoscopy team confirms readiness and continued until procedure completion. Administered only to participants in the Remifentanil Group.
  Other Names: Ultiva
  Arms: Remifentanil Group

SUMMARY:
This study compares two different sedation methods used during gastroscopy (a procedure to examine the upper digestive tract with a camera). Patients will be randomly assigned to receive either propofol-based sedation or remifentanil-based sedation, both combined with a standard premedication drug called midazolam.

During the procedure, the depth of sedation will be monitored using a device called a Bispectral Index (BIS) monitor, which measures brain activity to ensure patients receive the right amount of sedation-not too little and not too much. The sedation will be adjusted to keep patients comfortable but able to respond to simple commands.

The main goal of this study is to compare how quickly patients wake up after the procedure ends with each sedation method. The researchers will also measure:

* How quickly the procedure can begin after sedation starts
* How much sedation medication is needed
* How long the gastroscopy takes
* When patients are ready to go home
* Whether the BIS monitor readings match with clinical assessments of sedation
* Side effects such as low blood pressure, slow heart rate, or nausea
* How satisfied the endoscopist (the doctor performing the gastroscopy) is with the sedation quality

This research will help doctors understand which sedation approach provides better procedural efficiency, faster recovery, and fewer side effects for patients undergoing gastroscopy. Both propofol and remifentanil are already widely used and approved medications for sedation, and both will be given according to standard medical practice under careful monitoring.

Participants will be adults scheduled for routine diagnostic gastroscopy at Fatih Sultan Mehmet Training and Research Hospital. The study will enroll 80 patients total, with 40 patients in each sedation group.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE

Gastrointestinal endoscopy is one of the most commonly performed diagnostic procedures worldwide. Procedural sedation has become standard practice to enhance patient comfort, improve procedural quality, and increase patient willingness to undergo necessary endoscopic examinations.

Propofol is widely used for gastrointestinal endoscopy due to its rapid onset, predictable pharmacokinetics, and favorable recovery profile. However, propofol lacks intrinsic analgesic properties and may cause dose-dependent cardiovascular and respiratory depression, particularly when used as a sole agent.

Remifentanil is an ultra-short-acting opioid analgesic with context-insensitive pharmacokinetics, providing potent analgesia with rapid metabolism via plasma esterases. When combined with sedative agents, remifentanil may reduce hypnotic requirements and improve tolerance to endoscopic manipulation.

The Bispectral Index (BIS) is an electroencephalography-derived parameter that provides objective assessment of sedation depth. BIS values between 60 and 80 are conventionally targeted for moderate sedation. However, the clinical utility of BIS monitoring in gastrointestinal endoscopy and its correlation with clinical sedation scales remains incompletely characterized.

STUDY OBJECTIVES

Primary Objective:

To compare awakening time between propofol-based and remifentanil-based sedation regimens in patients undergoing diagnostic gastroscopy under BIS guidance.

Secondary Objectives:

1. To evaluate procedure start time (interval from sedation initiation to successful gastroscope insertion)
2. To assess total sedative consumption and procedure duration
3. To measure recovery characteristics and discharge time
4. To determine the correlation between BIS values and Ramsay Sedation Scale scores
5. To compare the incidence and severity of adverse events between groups
6. To evaluate endoscopist satisfaction with procedural conditions

STUDY DESIGN

This is a prospective, randomized, controlled, single-blind clinical trial. Patients will be randomized in a 1:1 ratio to receive either propofol-based or remifentanil-based sedation following midazolam premedication. Block randomization with variable block sizes will be used to ensure balanced allocation. Allocation concealment will be maintained using sequentially numbered, opaque, sealed envelopes.

Patients and outcome assessors will be blinded to group assignment. The anesthesiologist administering sedation will necessarily be unblinded to allow appropriate drug titration but will not participate in outcome assessment.

INTERVENTION DETAILS

All patients will receive:

* Standard monitoring: ECG, non-invasive blood pressure, pulse oximetry, BIS monitoring
* Supplemental oxygen via nasal cannula at 6 L/min
* Midazolam 2 mg intravenously as premedication

Group P (Propofol group):

Continuous propofol infusion at 100-150 µg/kg/min, titrated to maintain BIS 60-80 and Ramsay Sedation Scale 2-3.

Group R (Remifentanil group):

Remifentanil loading dose 1 µg/kg followed by continuous infusion at 0.025-0.1 µg/kg/min, titrated to maintain BIS 60-80 and Ramsay Sedation Scale 2-3.

OUTCOME MEASUREMENTS

Primary Outcome:

Awakening time, defined as time from cessation of sedative infusion to spontaneous eye opening in response to verbal command.

Key Secondary Outcomes:

* Procedure start time: Interval from sedation initiation to successful gastroscope insertion without patient movement or discomfort
* Total sedative drug consumption (mg for propofol, µg for remifentanil)
* Procedure duration (gastroscope insertion to withdrawal)
* Discharge time (Modified Aldrete Score ≥9)
* BIS-Ramsay correlation coefficient (Spearman's ρ)
* Adverse events: hypotension, bradycardia, desaturation, respiratory depression, postoperative nausea and vomiting
* Endoscopist satisfaction (5-point Likert scale)

Hemodynamic parameters (mean arterial pressure, heart rate, oxygen saturation), BIS values, and Ramsay Sedation Scale scores will be recorded at baseline and every 5 minutes throughout the procedure.

STATISTICAL ANALYSIS

Sample size calculation is based on the primary outcome (awakening time). Assuming mean awakening times of 5.0±2.0 minutes (propofol) versus 7.0±2.5 minutes (remifentanil), with α=0.05 and power=80%, a total of 80 patients (40 per group) will be required, accounting for 10% dropout.

Continuous variables will be compared using independent t-tests or Mann-Whitney U tests as appropriate. Categorical variables will be compared using chi-square or Fisher's exact tests. Repeated measures will be analyzed using ANOVA or GEE. BIS-Ramsay correlation will be evaluated using Spearman's rank correlation. Statistical significance is defined as p<0.05 (two-sided).

SAFETY CONSIDERATIONS

Both propofol and remifentanil are approved medications widely used for procedural sedation. All procedures will be performed by experienced personnel in a fully equipped endoscopy unit with immediate access to resuscitation equipment and medications. Adverse events will be managed according to standard clinical protocols and reported to the institutional ethics committee as required.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* ASA physical status I-III
* Scheduled for elective diagnostic gastroscopy
* Able to provide informed consent

Exclusion Criteria:

* ASA IV-V
* Pregnancy or lactation
* Known allergy to propofol, remifentanil, or midazolam
* Severe cardiopulmonary disease (NYHA III-IV, unstable angina, severe COPD requiring home oxygen)
* Chronic opioid use (>3 months daily use)
* BMI >40 kg/m²
* Obstructive sleep apnea requiring CPAP
* Severe hepatic or renal impairment
* Inability to provide informed consent
* Emergency procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-24 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Awakening Time | From end of procedure until awakening, assessed up to 30 minutes
  Time from cessation of sedative infusion (propofol or remifentanil) to spontaneous eye opening in response to verbal command ("Please open your eyes"). Measured in minutes.

SECONDARY OUTCOMES:
Total Sedative Drug Consumption | From sedation initiation to end of procedure, assessed up to 60 minutes
  Total amount of primary sedative agent administered during the procedure. Measured as total milligrams (mg) of propofol in the Propofol Group or total micrograms (µg) of remifentanil in the Remifentanil Group.

OTHER OUTCOMES:
Time to Discharge Readiness | From end of procedure until discharge readiness, assessed up to 2 hours
  Time from procedure completion to achievement of Modified Aldrete Score ≥9, indicating readiness for discharge from the endoscopy unit. The Modified Aldrete Score assesses activity, respiration, circulation, consciousness, and oxygen saturation (0-10 scale, ≥9 required for discharge). Measured in minutes.

CONTACTS AND LOCATIONS:
Overall Officials: cansu ofluoglu, md, Principal Investigator — Fatih Sultan Mehmet Training and Research Hospital, Department of Anesthesiology and Reanimation; doga meric yukselen, md, Study Director — Fatih Sultan Mehmet Training and Research Hospital, Department of Anesthesiology and Reanimation

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to protect participant privacy and confidentiality in accordance with local data protection regulations and institutional ethics committee requirements. Summary results will be published in peer-reviewed journals.